CLINICAL TRIAL: NCT04919655
Title: Clinical and Functional Expression Associated With CELSR1 Mutations in Primary Lymphedema of Lower Limbs
Brief Title: Primary Lymphedema and Mutation CELSR1 (Cadherin EGF LAG Seven-pass G-type Receptor 1)
Acronym: CELSR1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: GEHU - Duve Institute - Bruxelles (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0086
Record Dates: First submitted 2021-03-18; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Primary Lymphedema
Keywords: CELSR1; primary lymphedema of lower limbs; lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will describe the expression of mutation CELSR1 with codon stop and amino acids substitution mechanism in primary lymphedema, in both clinical examination and imaging exploration

DETAILED DESCRIPTION:
According to the literature, it seems that the mutation of the CELSR1 gene is associated with primary lymphedema.

Thus, the investigators have identified families with CELSR1 mutation with codon stop or animo acid substitution mechanisms among patients followed up in vascular medicine department, at Montpellier University hospital for primary lymphedema of lower limbs.

Among the mutation carriers, the investigators have collected the clinical examinations and imaging exploration results, realized systematically during the follow up of all the patient with primary lymphedema (venous Doppler, MRI of the lymphatic system, lymphoscintigraphy of the lower limbs, abdominal ultrasound), in order to search for a morphological and functional pattern associated with the mutation.

ELIGIBILITY:
Inclusion criteria:

* Patient followed up in vascular medicine departement at Montpellier University Hospital for primary lymphedema of lower limbs, who carries the CELSR1 mutation with codon stop or amino acids substitution mechanism.
* Relatives to the index case who carry the mutation for the segregation study.

Exclusion criteria:

* Patients who carry another mutation than CELSR1 responsible for primary lymphedema
* Syndromic form of primary lymphedema
* Patient not followed up at Montpellier University Hospital.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary lymphedema of lower limbs, which carriewho carry d the codon stop or the amino acids substitution CELSR1 mutation, followed up at Montpellier University Hospital regardless of the age.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Presence of unilateral lymphedema of lower limbs | day 1
  Describe the clinical examination of all CELSR1 mutation carriers: with ISL classification and perimeter measurement and Stemmer sign.
type of the morphological and functional pattern with imaging exploration. | day 1
  Describe the morphological and functional pattern of the CELSR1 mutation with the imaging exploration

SECONDARY OUTCOMES:
determine if deactivator mutation of CELSR1 | day 1
  determine if deactivator mutation of CELSR1 is associated with :
  * Great saphenous vein anatomical variation
  * kidney's anomalies

CONTACTS AND LOCATIONS:
Overall Officials: MESTRE GODIN Sandrine, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC